CLINICAL TRIAL: NCT00188708
Title: A Study of the Effect of Neoadjuvant Bicalutamide (Casodex) on Tumour Hypoxia in Patients With Clinically Localized Prostate Cancer
Brief Title: Effect of Casodex on Tumour Hypoxia - Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Trials Group (Network); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 00-0430-C; National Cancer Inst of Canada
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- hypoxia measurement (Experimental): Patients undergoing or planning to receive combined anti-androgen (Casodex) and radiotherapy
  Interventions: Procedure: hypoxia measurement

INTERVENTIONS:
Procedure: hypoxia measurement — transrectal oxygen measurement

SUMMARY:
Prostate cancers, in common with many other tumours, are often hypoxic; that is, they have low levels of oxygen. It is thought that tumour hypoxia may hasten the progression of cancers and make them more resistant to treatment. One previous study has suggested that hormone therapy, such as Casodex, may improve the prostate oxygen level. This study is designed to test that finding.

ELIGIBILITY:
Inclusion Criteria:

* Men with histologically proven prostatic carcinoma, stage cT2, N0, M0, receiving neoadjuvant bicalutamide plus conformal radiotherapy in study 9907, who have previously participated in the prostate cancer hypoxia project
* informed consent

Exclusion Criteria:

* Coagulopathy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-04; Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
To determine the effect of neoadjuvant anti-androgen therapy on oxygenation of prostatic tumours | 8 weeks
  Trans-rectal ultrasound and measurement of tumor oxygenation
Correlate level of tumor oxygenation with PSA level | 8 weeks
  PSA test (ug/L)
Correlate level of tumor oxygenation with hemoglobin level | 8 weeks
  hemoglobin test (g/L)
Correlate level of tumor oxygenation with prostate volume | 8 weeks
  prostate volume measurement

SECONDARY OUTCOMES:
To study of the effect of neoadjuvant anti-androgen therapy on prostate tumour histopathology and gene expression, and correlation of these effects with changes in oxygenation. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milosevic, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada